CLINICAL TRIAL: NCT03657251
Title: The MMRF CureCloud Multiple Myeloma Research Initiative
Brief Title: MMRF CureCloud Research Initiative
Status: Terminated | Type: Observational
Why Stopped: The MMRF has learned of the limitations of using a blood sample to collect genomic data, compared to a bone marrow aspirate. We decided that our resources are best served in other areas at this time.
Sponsor: Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MMRF-18-001
Record Dates: First submitted 2018-08-28; First posted 2018-09-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood will be collected from all participants after electronic online consenting via a mailed blood kit designed for a mobile phlebotomy appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CureCloud Direct to Patient
  Interventions: Genetic: liquid biopsy

INTERVENTIONS:
Genetic: liquid biopsy — Participants will be asked to provide up to a maximum total 40 mL of blood for all of the required sample collection. Peripheral blood will be collected from patients who consent to the protocol. These samples will be obtained at a time scheduled by the participant with the phlebotomy service provider, and will be collected at the participant's home. Patient peripheral blood samples can be obtained at diagnosis or at any time in follow up.

SUMMARY:
The MMRF CureCloud Research Initiative, a Direct-to-Patient Research effort aimed at enrolling 5,000 individuals from whom comprehensive molecular and immune analyses will be generated from blood specimens and the resulting data aggregated with the correlating clinical information. Blood will be collected from all participants after electronic online consenting via a mailed blood kit designed for a mobile phlebotomy appointment. Through the consenting process, participants will also be authorizing collection of their electronic medical records information.

DETAILED DESCRIPTION:
More than ever, there is an urgent need for a deeper understanding of the clinical, molecular and immune parameters involved in multiple myeloma disease initiation, progression and response to treatment. Such rich information, collected at the population level, is crucial to generate the evidence needed to ultimately make Precision Medicine a reality for all multiple myeloma patients. To this end the Multiple Myeloma Research Foundation (MMRF) is launching the MMRF CureCloud Research Initiative, a Direct-to-Patient Research effort aimed at enrolling 5,000 individuals from whom comprehensive molecular and immune analyses will be generated from blood specimens and the resulting data aggregated with the correlating clinical information. Blood will be collected from all participants after electronic online consenting via a mailed blood kit designed for a mobile phlebotomy appointment. Through the consenting process, participants will also allow the MMRF to collect their electronic medical records information. An important deliverable of the MMRF CureCloud Research Initiative is a curated dataset of integrated genomic, immune and correlating clinical data that will be made available to support scientific investigations through the MMRF CureCloud, a cloud-based platform with tools and capabilities for the seamless aggregation, integration and analysis of large collections of myeloma datasets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with active Multiple Myeloma
2. Patients have signed an online consent form

Exclusion Criteria:

1. Patients who live outside the United States
2. Patients with a diagnosis other than Multiple Myeloma or a known or suspected precursor to Multiple Myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol is designed to collect peripheral blood samples with annotated clinical data from patients with active Multiple Myeloma
Sampling Method: Probability Sample
Enrollment: 1105 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Collection and Analyses of Clinical Information and Peripheral Blood Samples | 5 years
  Patients that have been diagnosed with active Multiple Myeloma will be asked to share their clinical information and blood samples to help scientists and researchers understand these conditions better. The study will use submitted blood samples to perform comprehensive research that will include, among others, genomic and immune characterization, as well as collect past and present medical records to combine and compare with the blood sample analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hearn J Cho, MD, PhD, Principal Investigator — Multiple Myeloma Research Foundation; George Mulligan, PhD, Principal Investigator — Multiple Myeloma Research Foundation
Locations (4):
- United States (4):
  - Multiple Myeloma Research Foundation, Norwalk, Connecticut
  - Washington University Medical Campus, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Some data collected may be deposited into databases such as dbGAP and GDC. All identifiable information will be removed prior to submission so that the data cannot be linked to the participant in any way. The database of Genotypes and Phenotypes (dbGaP) and the he Genomic Data Commons (GDC) are databases developed by the National Cancer Institute (NCI) to archive and distribute the results of studies that have investigated the interaction of genotype and phenotype. Data submitted from this study to dbGAP and GDC will only be available through controlled access and restricted to cancer research studies. Any researcher requesting access to the data must formally apply and present a research study rationale for why they need access to the data. The data may also be submitted to other future database systems which will have similar access controls as dbGAP and GDC.